CLINICAL TRIAL: NCT01380730
Title: LAPLACE TIMI 57 - A Double-blind, Randomized, Placebo-controlled, Multicenter, Dose-ranging Study to Evaluate Tolerability and Efficacy of AMG 145 on LDL-C in Combination With HMG-CoA Reductase Inhibitors in Hypercholesterolemic Subjects
Brief Title: LAPLACE-TIMI 57: Low-density Lipoprotein Cholesterol (LDL-C) Assessment With PCSK9 monoclonaL Antibody Inhibition Combined With Statin thErapy
Acronym: LAPLACE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: The TIMI Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20101155
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Results first posted 2015-10-01 (Estimated); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Hyperlipidemia
Keywords: Hypercholesterolemia; Proprotein convertase subtilisin/kexin type 9 (PCSK9)
MeSH Terms: conditions — Hyperlipidemias; Hypercholesterolemia; Hypercholesterolemia, Autosomal Dominant, 3 | interventions — evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Placebo Q2W (Placebo Comparator): Participants received placebo subcutaneous injection once every 2 weeks (Q2W) for 12 weeks.
  Interventions: Other: Placebo to Evolocumab
- Placebo Q4W (Placebo Comparator): Participants received placebo subcutaneous injection once every 4 weeks (Q4W) for 12 weeks.
  Interventions: Other: Placebo to Evolocumab
- Evolocumab 70 mg Q2W (Experimental): Participants received 70 mg evolocumab by subcutaneous injection once every 2 weeks for 12 weeks.
  Interventions: Biological: Evolocumab
- Evolocumab 105 mg Q2W (Experimental): Participants received 105 mg evolocumab by subcutaneous injection once every 2 weeks for 12 weeks.
  Interventions: Biological: Evolocumab
- Evolocumab 140 mg Q2W (Experimental): Participants received 140 mg evolocumab by subcutaneous injection once every 2 weeks for 12 weeks.
  Interventions: Biological: Evolocumab
- Evolocumab 280 mg Q4W (Experimental): Participants received 280 mg evolocumab by subcutaneous injection once every 4 weeks for 12 weeks.
  Interventions: Biological: Evolocumab
- Evolocumab 350 mg Q4W (Experimental): Participants received 350 mg evolocumab by subcutaneous injection once every 4 weeks for 12 weeks.
  Interventions: Biological: Evolocumab
- Evolocumab 420 mg Q4W (Experimental): Participants received 420 mg evolocumab by subcutaneous injection once every 4 weeks for 12 weeks.
  Interventions: Biological: Evolocumab

INTERVENTIONS:
Biological: Evolocumab — Administered by subcutaneous injection
  Other Names: AMG 145; Repatha
  Arms: Evolocumab 105 mg Q2W; Evolocumab 140 mg Q2W; Evolocumab 280 mg Q4W; Evolocumab 350 mg Q4W; Evolocumab 420 mg Q4W; Evolocumab 70 mg Q2W
Other: Placebo to Evolocumab — Administered by subcutaneous injection
  Arms: Placebo Q2W; Placebo Q4W

SUMMARY:
To evaluate the effect of 12 weeks of subcutaneous (SC) evolocumab (AMG 145) administered every 2 weeks (Q2W) or every 4 weeks (Q4W), compared with placebo, on percent change from baseline in LDL-C when used in addition to a statin in adults with hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 to ≤ 80 years of age
* On an approved statin, with or without ezetimibe, with stable dose(s) for at least 4 weeks
* Fasting LDL-C ≥ 85 mg/dL
* Fasting triglycerides ≤ 400 mg/dL

Exclusion Criteria:

* Myocardial infarction, unstable angina, percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG) or stroke within 3 months prior to randomization
* Type 1 diabetes; newly diagnosed or poorly controlled type 2 diabetes (Glycosyated Hemoglobin (HbA1c) > 8.5%)
* Uncontrolled hypertension
* New York Heart Association (NYHA) III or IV heart failure, or known left ventricular ejection fraction < 30%
* Uncontrolled cardiac arrhythmia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 631 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2012-04-05 (Actual); Study Completion 2012-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (90):
- United States (51):
  - Research Site, Birmingham, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Malvern, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Carmichael, California
  - Research Site, Newport Beach, California
  - Research Site, Roseville, California
  - Research Site, Westlake Village, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Littleton, Colorado
  - Research Site, Daytona Beach, Florida
  - Research Site, Green Cove Springs, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Miami, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Peoria, Illinois
  - Research Site, Hammond, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, Iowa City, Iowa
  - Research Site, Lexington, Kentucky
  - Research Site, Auburn, Maine
  - Research Site, Bangor, Maine
  - Research Site, Portland, Maine
  - Research Site, Kalamazoo, Michigan
  - Research Site, Marquette, Michigan
  - Research Site, Ypsilanti, Michigan
  - Research Site, Tupelo, Mississippi
  - Research Site, Great Falls, Montana
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Cortlandt Manor, New York
  - Research Site, Williamsville, New York
  - Research Site, Smithfield, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Mansfield, Ohio
  - Research Site, Marion, Ohio
  - Research Site, Sandusky, Ohio
  - Research Site, Camp Hill, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, Florence, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Jackson, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Tacoma, Washington
  - Research Site, Madison, Wisconsin
- Canada (19):
  - Research Site, Burnaby, British Columbia
  - Research Site, Kelowna, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Cambridge, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Sarnia, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Woodstock, Ontario
  - Research Site, Gatineau, Quebec
  - Research Site, Lachine, Quebec
  - Research Site, Longueuil, Quebec
  - Research Site, Pointe-Claire, Quebec
  - Research Site, Québec, Quebec
- Czechia (7):
  - Research Site, Brno
  - Research Site, Olomouc
  - Research Site, Prague
  - Research Site, Slaný
  - Research Site, Svitavy
  - Research Site, Ústí nad Orlicí
  - Research Site, Znojmo
- Denmark (3):
  - Research Site, Aalborg
  - Research Site, Ballerup Municipality
  - Research Site, Vejle
- Hungary (10):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Dunaújváros
  - Research Site, Eger
  - Research Site, Gyula
  - Research Site, Kecskemét
  - Research Site, Komárom
  - Research Site, Mosonmagyaróvár
  - Research Site, Szolnok
  - Research Site, Zalaegerszeg

REFERENCES:
- [Background] Giugliano RP, Desai NR, Kohli P, Rogers WJ, Somaratne R, Huang F, Liu T, Mohanavelu S, Hoffman EB, McDonald ST, Abrahamsen TE, Wasserman SM, Scott R, Sabatine MS; LAPLACE-TIMI 57 Investigators. Efficacy, safety, and tolerability of a monoclonal antibody to proprotein convertase subtilisin/kexin type 9 in combination with a statin in patients with hypercholesterolaemia (LAPLACE-TIMI 57): a randomised, placebo-controlled, dose-ranging, phase 2 study. Lancet. 2012 Dec 8;380(9858):2007-17. doi: 10.1016/S0140-6736(12)61770-X. Epub 2012 Nov 6. PMID 23141813
- [Background] Kohli P, Desai NR, Giugliano RP, Kim JB, Somaratne R, Huang F, Knusel B, McDonald S, Abrahamsen T, Wasserman SM, Scott R, Sabatine MS. Design and rationale of the LAPLACE-TIMI 57 trial: a phase II, double-blind, placebo-controlled study of the efficacy and tolerability of a monoclonal antibody inhibitor of PCSK9 in subjects with hypercholesterolemia on background statin therapy. Clin Cardiol. 2012;35(7):385-91. doi: 10.1002/clc.22014. Epub 2012 Jun 19. PMID 22714699
- [Derived] Desai NR, Kohli P, Giugliano RP, O'Donoghue ML, Somaratne R, Zhou J, Hoffman EB, Huang F, Rogers WJ, Wasserman SM, Scott R, Sabatine MS. AMG145, a monoclonal antibody against proprotein convertase subtilisin kexin type 9, significantly reduces lipoprotein(a) in hypercholesterolemic patients receiving statin therapy: an analysis from the LDL-C Assessment with Proprotein Convertase Subtilisin Kexin Type 9 Monoclonal Antibody Inhibition Combined with Statin Therapy (LAPLACE)-Thrombolysis in Myocardial Infarction (TIMI) 57 trial. Circulation. 2013 Aug 27;128(9):962-9. doi: 10.1161/CIRCULATIONAHA.113.001969. Epub 2013 Jul 24. PMID 23884353
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled adults aged 18 - 80 years who were on a statin, with or without ezetimibe, with stable dose(s) for at least 4 weeks, and fasting low-density lipoprotein cholesterol (LDL-C) ≥ 85 mg/dL.
  The first patient enrolled on 18 July 2011 and the last patient enrolled on 22 December 2011.
Pre-assignment Details: Eligible participants were randomized equally into 1 of 8 treatment groups. Randomization was stratified by screening LDL-C level (< 130 mg/dL or ≥ 130 mg/dL) and ezetimibe use at baseline (yes or no).
Period: Overall Study
Arm/Group | Placebo Q2W | Placebo Q4W | Evolocumab 70 mg Q2W | Evolocumab 105 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 350 mg Q4W | Evolocumab 420 mg Q4W
Started | 78 | 79 | 79 | 79 | 78 | 79 | 79 | 80
Received Treatment | 78 | 77 (2 participants did not receive treatment but were followed until the end of study) | 79 | 79 | 78 | 79 | 79 | 80
Completed | 78 | 79 | 79 | 79 | 77 | 79 | 79 | 80
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (all randomized participants who received at least 1 dose of investigational product).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Q2W | Placebo Q4W | Evolocumab 70 mg Q2W | Evolocumab 105 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 350 mg Q4W | Evolocumab 420 mg Q4W | Total
Number analyzed (Participants) | 78 | 77 | 79 | 79 | 78 | 79 | 79 | 80 | 629
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (8.8) | 60.1 (9.6) | 59.4 (9.9) | 58.8 (9.7) | 62.4 (10.2) | 60.3 (8.4) | 61.9 (8.8) | 60.9 (10.3) | 60.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 41 | 44 | 25 | 45 | 40 | 38 | 44 | 319
  Male | 36 | 36 | 35 | 54 | 33 | 39 | 41 | 36 | 310
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 3
  Asian | 0 | 2 | 1 | 3 | 1 | 2 | 2 | 1 | 12
  Black or African American | 6 | 0 | 6 | 8 | 9 | 8 | 4 | 9 | 50
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 3
  White | 72 | 74 | 72 | 67 | 67 | 64 | 72 | 70 | 558
  Other | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 3
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 1 | 6 | 5 | 0 | 6 | 1 | 0 | 2 | 21
  Not Hispanic or Latino | 77 | 71 | 74 | 79 | 72 | 78 | 79 | 78 | 608
Stratification Factor: LDL-C Level [Number; unit: participants]
  < 130 mg/dL | 51 | 51 | 51 | 51 | 52 | 51 | 52 | 53 | 412
  ≥ 130 mg/dL | 27 | 26 | 28 | 28 | 26 | 28 | 27 | 27 | 217
Stratification Factor: Baseline Ezetimibe Use [Number; unit: participants]
  No | 71 | 69 | 72 | 72 | 71 | 72 | 72 | 73 | 572
  Yes | 7 | 8 | 7 | 7 | 7 | 7 | 7 | 7 | 57
LDL-C Concentration [Mean (Standard Deviation); unit: mg/dL] — LDL-C was measured using ultracentrifugation.
  mg/dL | 122.2 (27.1) | 124.9 (30.6) | 121.4 (24.4) | 127.4 (32.1) | 120.9 (25.1) | 122.0 (28.8) | 123.2 (27.1) | 120.8 (26.5) | 122.8 (27.7)
Non-High-Density Lipoprotein Cholesterol (non-HDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] | 146.9 (29.9) | 150.2 (36.5) | 145.3 (29.9) | 151.2 (37.2) | 145.3 (26.2) | 146.3 (33.3) | 150.0 (29.1) | 144.4 (31.2) | 147.4 (31.8)
Apolipoprotein B Concentration [Mean (Standard Deviation); unit: mg/dL] | 99.9 (17.0) | 101.6 (20.0) | 99.9 (16.8) | 103.6 (22.3) | 98.8 (16.6) | 101.3 (21.2) | 102.6 (18.9) | 99.9 (18.6) | 100.9 (19.0)
Total Cholesterol/HDL-C ratio [Mean (Standard Deviation); unit: ratio] | 3.940 (1.016) | 4.057 (1.303) | 4.002 (1.243) | 4.128 (1.473) | 3.932 (1.022) | 4.007 (1.300) | 4.118 (0.963) | 3.885 (1.090) | 4.008 (1.184)
Apolipoprotein B/Apolipoprotein A-1 Ratio [Mean (Standard Deviation); unit: ratio] | 0.660 (0.155) | 0.676 (0.194) | 0.675 (0.191) | 0.695 (0.219) | 0.649 (0.155) | 0.662 (0.199) | 0.687 (0.175) | 0.653 (0.177) | 0.670 (0.184)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at Week 12
Description: LDL-C was measured using ultracentrifugation.
Time Frame: Baseline and Week 12
Population: Full analysis set; missing ultracentrifugation LDL-C at Week 12 was imputed using last observation carried forward (LOCF) and calculated LDL-C.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo Q4W | Evolocumab 70 mg Q2W | Evolocumab 105 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 350 mg Q4W | Evolocumab 420 mg Q4W
Number analyzed (Participants) | 78 | 77 | 79 | 79 | 78 | 79 | 79 | 80
percent change | 2.76 (2.39) | -0.98 (2.51) | -39.06 (2.39) | -57.48 (2.39) | -63.34 (2.40) | -42.82 (2.52) | -50.98 (2.51) | -51.31 (2.53)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; The null hypothesis was that there was no mean difference in the percent change from Baseline at Week 12 in LDL-C between evolocumab and placebo, and the alternative hypothesis was that a mean difference did exist; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -66.10, 95% CI 2-sided [-71.48 to -60.72], Standard Error of Mean 2.73 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo Q2W vs Evolocumab 105 mg Q2W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -60.24, 95% CI 2-sided [-65.61 to -54.88], Standard Error of Mean 2.73 — Placebo is the reference
Statistical Analysis 3: Comparison: Placebo Q2W vs Evolocumab 70 mg Q2W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -41.82, 95% CI 2-sided [-47.18 to -36.45], Standard Error of Mean 2.73 — Placebo is the reference
Statistical Analysis 4: Comparison: Placebo Q4W vs Evolocumab 420 mg Q4W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -50.33, 95% CI 2-sided [-56.04 to -44.62], Standard Error of Mean 2.90 — Placebo is the reference
Statistical Analysis 5: Comparison: Placebo Q4W vs Evolocumab 350 mg Q4W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -50.00, 95% CI 2-sided [-55.69 to -44.31], Standard Error of Mean 2.89 — Placebo is the reference
Statistical Analysis 6: Comparison: Placebo Q4W vs Evolocumab 280 mg Q4W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — Multiplicity adjusted p-value is significant if less than the familywise error rate of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -41.84, 95% CI 2-sided [-47.55 to -36.13], Standard Error of Mean 2.90 — Placebo is the reference

2. Secondary Outcome: Change From Baseline in LDL-C at Week 12
Description: LDL-C was measured using ultracentrifugation.
Time Frame: Baseline and Week 12
Population: Full analysis set; missing data at Week 12 were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo Q2W | Placebo Q4W | Evolocumab 70 mg Q2W | Evolocumab 105 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 350 mg Q4W | Evolocumab 420 mg Q4W
Number analyzed (Participants) | 78 | 77 | 79 | 79 | 78 | 79 | 79 | 80
mg/dL | -0.2 (3.4) | -3.2 (3.3) | -50.9 (3.4) | -77.6 (3.5) | -79.5 (3.4) | -53.7 (3.3) | -64.3 (3.3) | -64.3 (3.3)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -79.2, 95% CI 2-sided [-87.0 to -71.5], Standard Error of Mean 4.0 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo Q2W vs Evolocumab 105 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -77.4, 95% CI 2-sided [-85.2 to -69.6], Standard Error of Mean 4.0 — Placebo is the reference
Statistical Analysis 3: Comparison: Placebo Q2W vs Evolocumab 70 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -50.7, 95% CI 2-sided [-58.5 to -43.0], Standard Error of Mean 4.0 — Placebo is the reference
Statistical Analysis 4: Comparison: Placebo Q4W vs Evolocumab 420 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -61.1, 95% CI 2-sided [-68.6 to -53.7], Standard Error of Mean 3.8 — Placebo is the reference
Statistical Analysis 5: Comparison: Placebo Q4W vs Evolocumab 350 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -61.1, 95% CI 2-sided [-68.5 to -53.7], Standard Error of Mean 3.8 — Placebo is the reference
Statistical Analysis 6: Comparison: Placebo Q4W vs Evolocumab 280 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -50.6, 95% CI 2-sided [-58.0 to -43.1], Standard Error of Mean 3.8 — Placebo is the reference

3. Secondary Outcome: Percent Change From Baseline in Non-High Density Lipoprotein Cholesterol (Non-HDL-C) at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set; missing data at Week 12 were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo Q4W | Evolocumab 70 mg Q2W | Evolocumab 105 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 350 mg Q4W | Evolocumab 420 mg Q4W
Number analyzed (Participants) | 78 | 77 | 79 | 79 | 78 | 79 | 79 | 80
percent change | 2.21 (2.20) | -1.26 (2.26) | -36.23 (2.20) | -53.21 (2.20) | -59.19 (2.21) | -39.05 (2.27) | -47.05 (2.26) | -48.83 (2.27)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -61.40, 95% CI 2-sided [-66.37 to -56.43], Standard Error of Mean 2.53 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo Q2W vs Evolocumab 105 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -55.42, 95% CI 2-sided [-60.37 to -50.47], Standard Error of Mean 2.52 — Placebo is the reference
Statistical Analysis 3: Comparison: Placebo Q2W vs Evolocumab 70 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -38.44, 95% CI 2-sided [-43.39 to -33.48], Standard Error of Mean 2.52 — Placebo is the reference
Statistical Analysis 4: Comparison: Placebo Q4W vs Evolocumab 420 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -47.58, 95% CI 2-sided [-52.72 to -42.44], Standard Error of Mean 2.61 — Placebo is the reference
Statistical Analysis 5: Comparison: Placebo Q4W vs Evolocumab 350 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -45.80, 95% CI 2-sided [-50.92 to -40.67], Standard Error of Mean 2.60 — Placebo is the reference
Statistical Analysis 6: Comparison: Placebo Q4W vs Evolocumab 280 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -37.79, 95% CI 2-sided [-42.94 to -32.65], Standard Error of Mean 2.61 — Placebo is the reference

4. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set; missing data at Week 12 were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo Q4W | Evolocumab 70 mg Q2W | Evolocumab 105 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 350 mg Q4W | Evolocumab 420 mg Q4W
Number analyzed (Participants) | 78 | 77 | 79 | 79 | 78 | 79 | 79 | 80
percent change | 5.86 (2.15) | 3.22 (2.25) | -28.88 (2.15) | -44.29 (2.14) | -50.59 (2.15) | -31.16 (2.26) | -37.55 (2.26) | -38.81 (2.27)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -56.45, 95% CI 2-sided [-61.28 to -51.61], Standard Error of Mean 2.46 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo Q2W vs Evolocumab 105 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -50.15, 95% CI 2-sided [-54.97 to -45.33], Standard Error of Mean 2.45 — Placebo is the reference
Statistical Analysis 3: Comparison: Placebo Q2W vs Evolocumab 70 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -34.74, 95% CI 2-sided [-39.56 to -29.92], Standard Error of Mean 2.45 — Placebo is the reference
Statistical Analysis 4: Comparison: Placebo Q4W vs Evolocumab 420 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -42.03, 95% CI 2-sided [-47.16 to -36.90], Standard Error of Mean 2.61 — Placebo is the reference
Statistical Analysis 5: Comparison: Placebo Q4W vs Evolocumab 350 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -40.77, 95% CI 2-sided [-45.88 to -35.66], Standard Error of Mean 2.60 — Placebo is the reference
Statistical Analysis 6: Comparison: Placebo Q4W vs Evolocumab 280 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -34.38, 95% CI 2-sided [-39.51 to -29.25], Standard Error of Mean 2.61 — Placebo is the reference

5. Secondary Outcome: Percent Change From Baseline in Total Cholesterol/HDL-C Ratio at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set; missing data at Week 12 were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo Q4W | Evolocumab 70 mg Q2W | Evolocumab 105 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 350 mg Q4W | Evolocumab 420 mg Q4W
Number analyzed (Participants) | 78 | 77 | 79 | 79 | 78 | 79 | 79 | 80
percent change | 2.64 (1.97) | -2.00 (1.90) | -28.76 (1.97) | -40.73 (1.97) | -45.09 (1.98) | -29.73 (1.91) | -37.97 (1.91) | -37.66 (1.92)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -47.74, 95% CI 2-sided [-52.18 to -43.29], Standard Error of Mean 2.26 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo Q2W vs Evolocumab 105 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -43.38, 95% CI 2-sided [-47.81 to -38.94], Standard Error of Mean 2.25 — Placebo is the reference
Statistical Analysis 3: Comparison: Placebo Q2W vs Evolocumab 70 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -31.40, 95% CI 2-sided [-35.83 to -26.97], Standard Error of Mean 2.25 — Placebo is the reference
Statistical Analysis 4: Comparison: Placebo Q4W vs Evolocumab 420 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -35.65, 95% CI 2-sided [-39.99 to -31.32], Standard Error of Mean 2.20 — Placebo is the reference
Statistical Analysis 5: Comparison: Placebo Q4W vs Evolocumab 350 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -35.97, 95% CI 2-sided [-40.29 to -31.65], Standard Error of Mean 2.20 — Placebo is the reference
Statistical Analysis 6: Comparison: Placebo Q4W vs Evolocumab 280 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -27.73, 95% CI 2-sided [-32.06 to -23.39], Standard Error of Mean 2.20 — Placebo is the reference

6. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B/Apolipoprotein A-1 Ratio at Week 12
Time Frame: Baseline and Week 12
Population: Full analysis set; missing data at Week 12 were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo Q2W | Placebo Q4W | Evolocumab 70 mg Q2W | Evolocumab 105 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 350 mg Q4W | Evolocumab 420 mg Q4W
Number analyzed (Participants) | 78 | 77 | 79 | 79 | 78 | 79 | 79 | 80
percent change | -0.30 (2.13) | -0.35 (2.38) | -35.04 (2.13) | -47.60 (2.12) | -53.73 (2.14) | -34.11 (2.40) | -42.74 (2.39) | -43.28 (2.40)
Statistical Analysis 1: Comparison: Placebo Q2W vs Evolocumab 140 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -53.44, 95% CI 2-sided [-58.23 to -48.65], Standard Error of Mean 2.44 — Placebo is the reference
Statistical Analysis 2: Comparison: Placebo Q2W vs Evolocumab 105 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -47.30, 95% CI 2-sided [-52.08 to -42.52], Standard Error of Mean 2.43 — Placebo is the reference
Statistical Analysis 3: Comparison: Placebo Q2W vs Evolocumab 70 mg Q2W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -34.75, 95% CI 2-sided [-39.53 to -29.97], Standard Error of Mean 2.43 — Placebo is the reference
Statistical Analysis 4: Comparison: Placebo Q4W vs Evolocumab 420 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -42.93, 95% CI 2-sided [-48.36 to -37.50], Standard Error of Mean 2.76 — Placebo is the reference
Statistical Analysis 5: Comparison: Placebo Q4W vs Evolocumab 350 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -42.40, 95% CI 2-sided [-47.81 to -36.98], Standard Error of Mean 2.75 — Placebo is the reference
Statistical Analysis 6: Comparison: Placebo Q4W vs Evolocumab 280 mg Q4W; Test type: Superiority or Other; p < 0.001, ANCOVA — Testing based on a significance level of 0.05; The ANCOVA model included treatment group and stratification factors; LS Mean Treatment Difference = -33.77, 95% CI 2-sided [-39.20 to -28.33], Standard Error of Mean 2.76 — Placebo is the reference

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo Q2W | Placebo Q4W | Evolocumab 70 mg Q2W | Evolocumab 105 mg Q2W | Evolocumab 140 mg Q2W | Evolocumab 280 mg Q4W | Evolocumab 350 mg Q4W | Evolocumab 420 mg Q4W
Serious Adverse Events (participants affected / at risk) | 4/78 | 0/77 | 0/79 | 1/79 | 4/78 | 2/79 | 2/79 | 2/80
Other Adverse Events (participants affected / at risk) | 15/78 | 17/77 | 20/79 | 28/79 | 27/78 | 21/79 | 23/79 | 30/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=78) | Placebo Q4W (N=77) | Evolocumab 70 mg Q2W (N=79) | Evolocumab 105 mg Q2W (N=79) | Evolocumab 140 mg Q2W (N=78) | Evolocumab 280 mg Q4W (N=79) | Evolocumab 350 mg Q4W (N=79) | Evolocumab 420 mg Q4W (N=80)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neurological symptom (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Substance abuse (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Penile haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Physical assault (Social circumstances) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Coronary artery bypass (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Q2W (N=78) | Placebo Q4W (N=77) | Evolocumab 70 mg Q2W (N=79) | Evolocumab 105 mg Q2W (N=79) | Evolocumab 140 mg Q2W (N=78) | Evolocumab 280 mg Q4W (N=79) | Evolocumab 350 mg Q4W (N=79) | Evolocumab 420 mg Q4W (N=80)
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 1 | 4 | 2 | 1 | 2 | 3
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 3 | 4 | 3 | 4
Fatigue (General disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 5
Influenza (Infections and infestations) | 2 | 1 | 3 | 3 | 6 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 6 | 5 | 9 | 8 | 7 | 8 | 8 | 8
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 2 | 3 | 4 | 0 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 4 | 5 | 2 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 2 | 4 | 3 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 1 | 1 | 1 | 4 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 4 | 1
Headache (Nervous system disorders) | 2 | 0 | 1 | 1 | 4 | 1 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 3 | 0 | 6 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.